CLINICAL TRIAL: NCT06738680
Title: PRedictive Value of Multiparametric Dynamic Whole-body 18F-FDG-PET Imaging on a LAFOV System for FIRST-line Chemo-immunotherapy Efficacy in Advanced Non-small-cell Lung Cancer: PROFIL-1 Study
Brief Title: PRedictive Value of Multiparametric Dynamic WB 18F-FDG-PET Imaging on a LAFOV System for FIRST-line Chemo-immunotherapy Efficacy in Advanced Non-small-cell Lung Cancer: PROFIL-1
Acronym: PROFIL-1
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0049
Record Dates: First submitted 2024-11-15; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Chemo-immunotherapy; Non-Small Cell Lung Cancer; Metastatic; Imaging Biomarkers; Prediction of response
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Radionuclide Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: LAFOV system (an innovative, latest-generation system) scan — To collect data from the LAFOV system (an innovative, latest-generation system) during the PET scan planned as part of your treatment.

SUMMARY:
Lung cancer is the leading cause of cancer deaths worldwide. Revolution of chemo-immunotherapy (CT-IO) in first-line of metastatic non-small-cell lung cancers (NSCLC) without actionable genomic alterations (AGAs) has dramatically improved prognosis, providing long response to a subset of patients. Because of a highly heterogeneous disease, majority of patients do not show long term benefit. Long axial field of view positron emission tomography (LAFOV-PET) scanner is a new emerging system allowing dynamic whole-body imaging with higher sensitivity, representing unique opportunity for oncological applications. The aim of this study is to determine if LAFOV-PET imaging biomarkers could early predict response to CT-IO in NSCLC.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer deaths worldwide. Revolution of chemo-immunotherapy (CT-IO) in first-line of metastatic non-small-cell lung cancers (NSCLC) without actionable genomic alterations (AGAs) has dramatically improved prognosis, providing long response to a subset of patients. Because of a highly heterogeneous disease, majority of patients do not show long term benefit. Long axial field of view positron emission tomography (LAFOV-PET) scanner is a new emerging system allowing dynamic whole-body imaging with higher sensitivity, representing unique opportunity for oncological applications. The aim of this study is to determine if LAFOV-PET imaging biomarkers could early predict response to CT-IO in NSCLC.

PROFIL-1 is a multicentre, single-arm, prospective non-interventional pilot study investigating the predictive value of multiparametric 18F-fluoro-deoxyglucose whole-body dynamic PET imaging on a LAFOV system for first-line CT-IO efficacy in advanced NSCLC, with a planned enrolment of 120 patients at 2 French sites. Adult patients with treatment-naïve advanced non-squamous or squamous NSCLC without AGAs and eligible for first-line CT-IO will be recruited for PROFIL-1. Patients will undergo LAFOV-PET before and after CT-IO induction. The primary objective is to evaluate predictive performance of a whole-body multiparametric analysis (radiomics and dynamics) in LAFOV-PET on CT-IO efficacy based on progression-free survival (PFS) per RECIST v1.1 by investigators. Secondary endpoints included correlations between imaging parameters and clinico-pathological characteristics, comparison between direct Patlak and indirect Patlak methods to determine dynamic parameters such as Ki (the net influx rate) and distribution volume (DV), number of tumor lesions and signal-to-noise ratio, objective response rate (ORR), overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years
* With advanced, non-operable, non-radiatable or metastatic NSCLC
* Treatment-naïve patients
* Eligible for first-line chemo-immunotherapy (anti-PD-1)
* Written Non-objection
* Eligible for LAFOV FDG-PET less than 21 days before initiation of treatment

Exclusion Criteria:

* Minor patients <18 years
* Oncogenic addiction targetable in 1st line: EGFR, ALK, ROS1, RET
* Pregnancy or breast-feeding
* Other histology than NSCLC
* Ineligible for first-line chemo-immunotherapy
* PET-FDG Scan contraindications
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable locally advanced non-irradiable or metastatic NSCLC, whose files are presented to the thoracic oncology Multidisciplinary Team at the Brest University Hospital and the Morlaix University Hospital, and for whom chemo-immunotherapy is indicated as 1st line treatment.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
1-year Progression-Free Survival | From date of chemo-immunotherapy initiation until the date of first documented progression or date of death, assessed up to 100 months.
  The primary endpoint is 1-year Progression-Free Survival (PFS) rate. PFS is defined as the time from chemo-immunotherapy initiation to the date of the first documented event of tumor progression or death in the absence of disease progression, whichever came first, assessed up to 100 months.

SECONDARY OUTCOMES:
Measurement of Ki images | From baseline PET/CT before chemo immunotherapy in ml/min/100 g
  Measurement of Ki images PET/CT parameters based on direct and indirect Patlak reconstruction methods with PBIF or IDIF in LAFOV-PET from baseline PET/CT before chemo immunotherapy
Measurement of distribution volume | From baseline PET/CT before chemo immunotherapy in L/kg
  Measurement of distribution volume dynamic PET/CT parameter based on direct and indirect Patlak reconstruction methods with PBIF or IDIF in LAFOV-PET from baseline PET/CT before chemo immunotherapy
Correlation between quantitative dynamic and radiomic parameters and clinico-histopathological parameters | From baseline PET/CT before chemo immunotherapy
  Correlation analyses between quantitative dynamic and radiomic PET derived parameters and clinico-histopathological parameters (clinical, biology, histology, genomic).
Contrast-to-noise ratio (CNR) | From baseline LAFOV PET/CT
  Contrast-to-noise ratio (CNR) (indicating the image quality in the lesion)
Target-to-background ratio (TBR) | From baseline LAFOV PET/CT
  Target-to-background ratio (TBR), defined as the ratio of the lesions' SUVmax and the SUVmean of healthy liver tissue (background) determined for each reconstruction algorithm
Objective response rate (ORR) | From baseline LAFOV PET to end of 1 year of treatment
  Objective response rate (ORR), defined as the proportion of patients experiencing an objective response (either complete response [CR] or partial response [PR]) as best response to CT-IO according to RECIST 1.1 criteria
Metabolic response rate (MRR) | From baseline LAFOV PET to end of 1 year of treatment
  Metabolic response rate (MRR), defined as the proportion of patients experiencing a metabolic response (either complete metabolic response [CMR] or partial metabolic response [PMR]) as best response to CT-IO according to Positron Emission Tomography Response Criteria in Solid Tumors version 1.0 (PERCIST v1.0)
Overall Survival | From date of chemo-immunotherapy initiation until the date of death from any cause, assessed up to 100 months
  Overall Survival, defined as the time from chemo-immunotherapy initiation until the date of death from any cause, assessed up to 100 months
Safety | From baseline LAFOV PET to end of 1 year of treatment
  Safety and tolerability according to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0.; Patient reported outcomes according to EQ-5D-5L and EORTC QLQ-C30 (baseline, 3 months, 6 months, 12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Margaux GEIER, Study Director — University Hospital, Brest
Locations (2):
- France (2):
  - Brest University Hospital, Brest
  - Morlaix Hospital Center, Morlaix

IPD SHARING:
Plan to Share IPD: Undecided